CLINICAL TRIAL: NCT04299360
Title: Comparison of Multi-point Pacing and Conventional CRT Through Non-invasive Hemodynamics Measurement and Global Longitudinal Strain Assessment
Acronym: COMPACT-MPP
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Universitaria Mater Domini, Catanzaro (Other)
Responsible Party: Principal Investigator, Antonio Curcio, Associate professor of Cardiology, Azienda Ospedaliera Universitaria Mater Domini, Catanzaro
Other Study IDs: 178
Record Dates: First submitted 2018-07-12; First posted 2020-03-06 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Cardiac Resynchronization Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- standard BIV: the following group describes the effects of the left ventricular stimulation involving a dipole of two electrodes located inside a suitable vessel branch of the coronary sinus (CS). Standard BIV pacing modality can be achieved by either a quadripolar electrode implanted in the CS, of which only two poles will be used for cardiac resynchronization therapy, or by a bipolar electrode equipped with just two electrodes. The latter describes the old technology, requiring a change into typology of generator which has to display an IS-1 connection (due to different distal terminal of the electrode itself), instead of the new one IS-4 connection that has been developed for quadripolar electrodes.
- MPP BIV: Such modality of left ventricular stimulation requires a dynamic use of the four electrodes located in the proximal segment of the electrocatheter that allows the recruitment of a vast area of the left ventricle. It is limited by the presence of scars on left ventricle surface, or phrenic nerve inadvertent stimulation.
  Interventions: Device: Cardiac Resynchronization Therapy device programming

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy device programming — Implanted CRT-D devices settings will be programmed based on the best acute hemodynamic response assessed non-invasively
  Groups: MPP BIV

SUMMARY:
Pilot, perspective, multi-center non-randomized study comparing Multi-point pacing and conventional CRT through non-invasive hemodynamics measurement and Global Longitudinal Strain assessment

ELIGIBILITY:
Inclusion Criteria:

* Recent or scheduled implantation of CRT-D system with quadripolar lead and MPP technology in patient with indications to CRT according to current guidelines

Exclusion Criteria:

* Patients in Atrial Tachycardia (AT) or Atrial Fibrillation (AF) at the time of the enrollment or with persistent or long-standing persistent/chronic AF
* NYHA IV patients
* Right Bundle Branch Block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Patients with standard indications to CRT satisfying the study Inclusion and Exclusion Criteria
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Acute improvement in cardiac function (1) | 24-48 hours after CRT-D implantation
  change in dP/dtmax, expressed in mmHg/s, assessed through photoplethysmography. This assessment represents in a non-invasive fashion, the rise in pressure (P) developed inside left ventricle during contraction over time.
Acute improvement in cardiac function (2) | 24-48 hours after CRT-D implantation
  change in global longitudinal strain, assessed through echocardiography. This assessment elucidates longitudinal shortening of the left ventricle as a percentage (change in length as a proportion to baseline length). GLS is derived from speckle tracking, and analyzed by post-processing of apical images of the left ventricle.

SECONDARY OUTCOMES:
Delayed response (1) | 3 Months
  change in GLS. Participants will investigate whether left ventricular remodeling upon "patient-tailored" biventricular stimulation will behave differentially according to type of stimulation; the total amount of CRT-responder patients will be therefore considered
Delayed response (2) | 3 Months
  change in NYHA class. Participants will check if functional status will change after optimized biventricular stimulation therapy and will provide clinical data on CRT responders.

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Azienda Ospedaliera Policlinico Mater Domini, Catanzaro, CZ
  - AO Cardarelli, Napoli
  - AOU Federico II, Napoli

REFERENCES:
- [Derived] Passafaro F, Rapacciuolo A, Ruocco A, Ammirati G, Crispo S, Pasceri E, Santarpia G, Mauro C, Esposito G, Indolfi C, Curcio A. COMPArison of Multi-Point Pacing and ConvenTional Cardiac Resynchronization Therapy Through Noninvasive Hemodynamics Measurement: Short- and Long-Term Results of the COMPACT-MPP Study. Am J Cardiol. 2024 Mar 15;215:42-49. doi: 10.1016/j.amjcard.2023.12.057. Epub 2024 Jan 17. PMID 38237796